CLINICAL TRIAL: NCT05060068
Title: Effect of Intravenous S-ketamine on Opioid Consumption and Postoperative Pain in Patients Undergoing Breast Cancer Surgery：a Multicenter, Randomised, Control Trial
Brief Title: Effect of Intravenous S-ketamine on Opioid Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yun Wu, Principal Investigator, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YX2021-070(F1)
Record Dates: First submitted 2021-08-22; First posted 2021-09-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Surgery
Keywords: breast cancer surgery; S-ketamine; opioid consumption
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The syringes and infusions will be identical for all of the groups and will run at the same rate in all subjects to enable blinding of the investigators. Outcomes will be evaluated by anesthesiologists who are blinded to the treatment allocation. Patients, nurses, observers, and the statistician will be blinded to patient allocation throughout the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo group (Placebo Comparator): Patients in the placebo group will receive a bolus of 0.9% saline, followed by continuous infusion of 0.9% saline until 30 min prior to the end of the surgery.
  Interventions: Drug: Placebo
- Low-dose ketamine group (Experimental): Patients in the low-dose ketamine group will receive a bolus of 0.5 mg/kg S-ketamine in saline, followed by continuous infusion of 2 μg/kg/min S-ketamine in saline until 30 min prior to the end of the surgery.
  Interventions: Drug: S-ketamine (low dose)
- High-dose ketamine group (Experimental): Patients in the low-dose ketamine group will receive a bolus of 0.5 mg/kg S-ketamine in saline, followed by continuous infusion of 4 μg/kg/min S-ketamine in saline until 30 min prior to the end of the surgery.
  Interventions: Drug: S-ketamine (high dose)

INTERVENTIONS:
Drug: S-ketamine (low dose) — Patients in the low-dose ketamine group will receive a bolus of 0.5 mg/kg S-ketamine in saline, followed by continuous infusion of 2 μg/kg/min S-ketamine in saline until 30 min prior to the end of the surgery.
  Other Names: LKET
  Arms: Low-dose ketamine group
Drug: Placebo — Patients in the placebo group will receive a bolus of 0.9% saline, followed by continuous infusion of 0.9% saline until 30 min prior to the end of the surgery.
  Other Names: CON
  Arms: Placebo group
Drug: S-ketamine (high dose) — Patients in the high-dose ketamine group will receive a bolus of 0.5 mg/kg S-ketamine in saline, followed by continuous infusion of 4 μg/kg/min S-ketamine in saline until 30 min prior to the end of the surgery.
  Other Names: HKET
  Arms: High-dose ketamine group

SUMMARY:
Female patients with an American Society of Anesthesia (ASA) physical status I-II, scheduled for elective breast cancer surgery will be included in the study. Subjects will be randomly assigned to one of three groups: the placebo group, the low-dose S-ketamine group, and the high-dose S-ketamine group. The primary outcome is the consumption of sufentanil during the surgery.

DETAILED DESCRIPTION:
All patients will be scheduled to a propofol-remifentanil general anesthesia and receive non-steroid anti-inflammatory drug before incision. Bolus sufentanil will be administered according to the blood pressure, heart rate and bispectral index perioperatively. Patients unable to understand the study procedure or unable to give informed consent, with concurrent analgesic or sedative medication, with history of chronic pain, psychiatric disorders, or alcohol or drug abuse, with an allergy to the study medication, who are pregnant or breast feeding, with a BMI >30 and <18 kg/m2, with severe cardiac, pulmonary, hepatic or renal dysfunction, with intracranial hypertension will be excluded.

Subjects will be randomly assigned to one of three groups: the placebo group, the low-dose S-ketamine group, and the high-dose S-ketamine group. The study medication will be administered in a bolus injected over 30 s after induction, followed by continuous infusion, which started after the initial bolus. The placebo group will receive a bolus of 0.9% saline, followed by continuous infusion of 0.9% saline. The low-dose ketamine group will be administered a bolus of 0.5 mg/kg S-ketamine in saline, followed by 2μg/kg/min S-ketamine in saline, whereas the high-dose ketamine group will be administered a bolus of 0.5 mg/kg S-ketamine in saline, followed by continuous infusion of 4μg/kg/min S-ketamine in saline. The syringes and infusions will be identical for all of the groups and will run at the same rate in all subjects to enable blinding of the investigators. Study medication will be terminated 30 min prior to the end of the surgery. After surgery and in the postanesthesia care unit, patients will be asked about their pain level on a numeric rating scale (NRS), and about the presence of intraoperative awareness, nausea, vomiting, and hallucinations. Rescue analgesia of sufentanil will be provided when NRS ≥ 4 or patients require. Pain level will also be assessed at 0.5, 2, 4, 6, 12 and 24 hour postoperatively as well as 3 and 6 month after the surgery. Depression scale will be evaluated before the surgery and in the 7th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with an American Society of Anesthesia (ASA) physical status I-II
2. Scheduled for elective breast cancer surgery

Exclusion Criteria:

1. Patients unable to understand the study procedure or unable to give informed consent
2. with concurrent analgesic or sedative medication,
3. with history of chronic pain
4. with history of psychiatric disorders
5. with history of alcohol or drug abuse
6. with an allergy to the study medication
7. who are pregnant or breast feeding
8. with a BMI >30 and <18 kg/m^2
9. with severe cardiac, pulmonary, hepatic or renal dysfunction
10. with intracranial hypertension

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
consumption of sufentanil | during the surgery
  the consumption of sufentanil during the surgery.

SECONDARY OUTCOMES:
postoperative pain assessment | at 0.5, 2, 4, 6, 12 and 24 hours respectively after surgery; Month 3 and Month 6 after surgery
  Patients will be asked about their pain level at rest and moving on a numeric rating scale evaluated on a 11-point (0 = no pain, 10 = worst pain imaginable).
consumption of analgesics | in the first 24 hour after surgery
  cumulative analgesic consumption after surgery
Richmond Agitation-Sedation Scale (RASS) | 30 minutes after surgery
  Richmond Agitation-Sedation Scale is a 10-point scale. The values and definitions for each level of agitation and sedation are displayed as follows: +4, Combative, overtly combative or violent; immediate danger to staff; +3, Very agitation, pulls on or removes tube(s) or catheter(s) or has aggressive behavior toward staff; +2, Agitated, frequent nonpurposeful movement or patient-ventilator dyssynchrony; +1, Restless, anxious or apprehensive but movements not aggressive or vigorous; 0, Alert and calm; -1, Drowsy, not fully alert, but has sustained (more than 10 seconds) awakening, with eye contact, to voice; -2, Light sedation, briefly (less than 10 seconds) awakens with eye contact to voice; -3, Moderate sedation, any movement (but no eye contact) to voice; -4, Deep sedation, no response to voice, but any movement to physical stimulation; -5, Unarousable, no response to voice or physical stimulation
sleep quality scale | sleep quality scale will be assessed in the morning (8:00 am）of first postoperative day
  Quality of sleep in the night of surgery day using a 4-point scale (1 = "slept well," 2 = "disturbed sleep," 3 = "nightmares," and 4 = "sleepless") will be recorded.
consumption of propofol | during the surgery
  the consumption of propofol during the surgery.
consumption of remifentanil | during the surgery
  the consumption of remifentanil during the surgery.
length of anesthesia | at the end of anesthesia
  from beginning to the end of anesthesia
length of surgery | at the end of surgery
  from beginning to the end of surgery
recovery time | at the time when patients waking up
  awakening time from surgery
consumption of vasoactive agents | during the surgery
  the consumption of any vasoactive agent (such as phenylephrine, urapidil, ephedrine)
blood pressure | before anesthesia, prior to incision, 5, 10, 30, 60 and 120 minutes after incision, at the end of surgery and 30 minutes after surgery
  noninvasive blood pressure
heart rate | before anesthesia, prior to incision, 5, 10, 30, 60 and 120 minutes after incision, at the end of surgery and 30 minutes after surgery
  Heart rate of the patients
bispectral index | before anesthesia, prior to incision, 5, 10, 30, 60 and 120 minutes after incision, at the end of surgery and 30 minutes after surgery
  Bispectral index during the surgery
adverse effects | through 24 hours after the surgery
  The presence of intraoperative awareness, nausea, vomiting, and hallucinations after surgery
Edinburgh postnatal depression scale | before surgery, at the 7th day and 3 months after surgery
  Depression scale generated from Edinburgh postnatal depression scale will be assessed. The minimum value is 0, and the maximum value is 30. The higher score means the higher possibility of depression.
ambulation time | 7 days after surgery
  interval time of patients' transit from bed rest to ambulation after surgery
hospitalization postoperatively | two weeks after surgery
  days of hospital staying after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, M.D., Ph. D., Study Chair — The Second Hospital of Anhui Medical University
Locations (1):
- Second Affiliated Hospital of Anhui Medical University, Hefei, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will become available when summary data are published.
Access Criteria: Yun Wu and Ye Zhang will review requests and criteria to share IPD. Requests are to be sent by email to wuyunanyi@163.com or zhangye_hassan@sina.com.

REFERENCES:
- [Background] Brinck ECV, Maisniemi K, Kankare J, Tielinen L, Tarkkila P, Kontinen VK. Analgesic Effect of Intraoperative Intravenous S-Ketamine in Opioid-Naive Patients After Major Lumbar Fusion Surgery Is Temporary and Not Dose-Dependent: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Anesth Analg. 2021 Jan;132(1):69-79. doi: 10.1213/ANE.0000000000004729. PMID 32167978
- [Background] Hamp T, Baron-Stefaniak J, Krammel M, Reiter B, Langauer A, Stimpfl T, Plochl W. Effect of intravenous S-ketamine on the MAC of sevoflurane: a randomised, placebo-controlled, double-blinded clinical trial. Br J Anaesth. 2018 Dec;121(6):1242-1248. doi: 10.1016/j.bja.2018.08.023. Epub 2018 Oct 15. PMID 30442251